CLINICAL TRIAL: NCT03289663
Title: Effectiveness Study of Bednets Treated With Synegistic Combination of Insectcides in an Area With Pyrethroid-resistant Vectors in the Democratic Republic of the Congo
Brief Title: Effectiveness Study of New Generation Bednets in the Context of Conventional Insecticide Resistance in the Democratic Republic of the Congo
Acronym: Net-PBO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université de Lubumbashi (Other)
Collaborators: Universiteit Antwerpen (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gillon Ilombe Kaounga, Researcher, Ministry of Public Health, Democratic Republic of the Congo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NET-06-08-76
Record Dates: First submitted 2017-08-10; First posted 2017-09-21 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Insecticide Resistance
Keywords: synergistic combination; insecticide resistance; vectors
MeSH Terms: interventions — Pyrethrins

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial
Who Masked: Participant
Masking Description: The 2 groups of villages will randomly receive either the bednets treated with conventional insecticide (Pyrethroid) or the synergistic combination of insecticides. None of the groups knows which bednets they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): The arm will receive bednets treated with conventional insecticide (Pyrethroid)
  Interventions: Drug: Pyrethroids
- Experimental (Experimental): The arm will receive bednets treated with new generation of insecticides (synergistic combination of insecticides)
  Interventions: Drug: synergistic combination of insecticides

INTERVENTIONS:
Drug: synergistic combination of insecticides — third generation insecticide -treated bednets
  Arms: Experimental
Drug: Pyrethroids — Conventional insecticide
  Arms: Control

SUMMARY:
Despite the mass distribution of LLINs (long-lasting insecticidal nets) as a Malaria control strategy, populations are still continuously exposed to a high frequency of malarial inoculation in some countries. The situation can be explained by a swift increase in the resistance of Anopheles to common insecticides. To preserve the gains of insecticides and improve their effectiveness, a new generation of bednets treated with piperonyl butoxide combination insectides have emerged.But more evidence is needed to plead for scale up of their usage. The lack of information relating to the additional impact of that combination on the transmission of Malaria, its relative efficacy in real-life setting and its safety in users are the rationale for more investigation.This will be a randomized controlled study on a dynamic cohort of households with 1680, 0-10 years-old subjects in 30 villages will be recruited to compute the effectiveness of this new tool.

The findings will be useful information for decision-making by national malaria control programs, their partners, the international community and the bednet manufacturers with regard to the effectiveness of the new combination of insecticides in real-life context. The results will also enable a better design of the tool in the future and a broader understanding of long-term dynamics for sustainability, as well as identification of some factors with negative impacts on the benefits of the strategy.

ELIGIBILITY:
Inclusion Criteria : -households where there are one or more children below the age of 10 years;

* Ability and willingness of the head of the household to participate based on signed informed consent (or fingerprint) and with the assistance of an impartial witness (if the head of the household is illiterate)

Exclusion Criteria :

* refusal of the head of household to participate
* known allergy to insecticides

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1680 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of laboratory confirmed clinical cases of Malaria | Participants will be actively followed up for 12 months. And any suspected case of clinical Malaria will immediately lead to microscopy and RDT for confirmation
  Microscopy to confirm the diagnosis of Malaria
Sporozoite rate | Anopheles mosquitoes will be captured every 3 months during 1 year
  Sporozoite detection by ELISA to determine infectivity of anopheles

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Général de Référence Saint Luc, Kisantu, Bas-Congo Province, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gleave K, Lissenden N, Chaplin M, Choi L, Ranson H. Piperonyl butoxide (PBO) combined with pyrethroids in insecticide-treated nets to prevent malaria in Africa. Cochrane Database Syst Rev. 2021 May 24;5(5):CD012776. doi: 10.1002/14651858.CD012776.pub3. PMID 34027998